CLINICAL TRIAL: NCT03187275
Title: Efficacy of Massage for the Treatment of Cancer-Related Fatigue (CRF) in Prostate Cancer Survivors
Acronym: mProstate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Mark H. Rapaport, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00095260
Record Dates: First submitted 2017-06-13; First posted 2017-06-14 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Cancer-related Problem/Condition
Keywords: Cancer Related Fatigue (CRF); Prostate Cancer; Swedish Massage Therapy (SMT); Cancer; Quality of Life (QOL)
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swedish Massage Therapy (Experimental): Participants in this arm will receive Swedish massage, which is the most commonly offered and best-known type of massage.
  Interventions: Other: Swedish Massage Therapy
- Light Touch Intervention (Active Comparator): Participants in this arm will receive light touch only.
  Interventions: Other: Light Touch Intervention

INTERVENTIONS:
Other: Swedish Massage Therapy — The therapist uses non-aromatic massage oil to facilitate making long, smooth strokes over the body. Swedish massage is done with the subject covered by a sheet, a technique called "draping." One part of the body is uncovered, massaged, and then covered up before moving onto another part of the body. Primary techniques used in the research protocol therapy are: effleurage, petrissage, tapotement. These will be administered according to a very specific, standardized protocol. The total session time will be 45 minutes.
  Other Names: SMT
  Arms: Swedish Massage Therapy
Other: Light Touch Intervention — The light-touch research intervention is based on the concept that there will be a noticeable effect with regard to massage when compared to light-touch alone without the massage. The protocol followed will be the same as the massage protocol other than that the therapist will use light-touch only. The total session time will be 45 minutes.
  Other Names: LT
  Arms: Light Touch Intervention

SUMMARY:
Cancer-related fatigue (CRF) is a prevalent and debilitating symptom experienced by cancer survivors. CRF can persist for months or years after cancer therapy is completed and has a negative impact on all areas of mental and physical function. Treatment options for CRF are extremely limited and finding safe, inexpensive, and effective interventions for managing this distressing symptom are urgently needed. Massage therapy is one of the fastest growing complementary therapies. A recently completed study in breast cancer survivors with CRF found that Swedish Massage Therapy (SMT) caused a significant reduction in fatigue and improvement in quality of life. This study investigates the effects of massage therapy on CRF among prostate cancer survivors. The study will evaluate whether SMT improves quality of life, depression, and anxiety. Second, this study will evaluate if SMT reduces CRF by decreasing the pro-inflammatory cytokine Interleukin-6 (IL-6). Lastly, to establish measures of reduced fatigue beyond self report at the treatment visits, the researchers will implement continuous, real-time monitoring of physiologic and psychological signs and symptoms, throughout the treatment period. This study will improve care for CRF and other hard-to-manage symptoms of cancer treatment and provide preliminary evidence of immune modulation as a potential mechanism of action.

This study is a randomized clinical trial to test the efficacy of Swedish massage therapy (SMT) versus an active control condition (light touch, LT) on cancer related fatigue in men with prostatic cancer, at least 2 months after the end of their radiation therapy. The primary outcome is the Multidimensional Fatigue Inventory (MFI). Secondary outcomes are the Patient-Reported Outcomes Measurement System (PROMIS) Fatigue Scale, plasma concentrations of cytokine IL-6, self-reported quality of life, depression, and anxiety, wearable measures of activity and sleep, and Automated Monitoring of Symptom Severity (AMoSS) ratings.

DETAILED DESCRIPTION:
Fatigue is the most common, and one of the most devastating symptoms among patients with cancer. According to the National Comprehensive Cancer Network (NCCN), cancer-related fatigue (CRF) is "a distressing, persistent, subjective sense of physical, emotional, and/or cognitive exhaustion related to cancer or its treatment that is not proportional to recent activity". Fatigue occurs across the spectrum of cancer types and treatments. CRF has a negative impact on all areas of function, including mood, physical function, work performance, social interaction, family care, cognitive performance, schoolwork, and community activities. CRF has been rated as more troublesome and to have a greater negative impact on quality of life than other cancer-related symptoms such as pain, depression, and nausea. CRF can persist for months or years after cancer therapy is completed.

Meaningful, evidence-based treatment options for CRF are limited. Over 50% of patients with cancer have used a complementary and alternative medicine (CAM) approach for symptom management and quality of life. One of the widely employed CAM interventions is massage therapy. Most of the studies investigating massage for patients with cancer focus on depression, anxiety, or pain as the outcomes of interest. A previous investigation of breast cancer survivors reported decreases in mood symptoms and an improvement in fatigue, however, CRF was not the primary outcome measure. This randomized clinical trial will test the efficacy of Swedish massage therapy (SMT) vs. an active control condition (light touch, LT) on cancer related fatigue in men with prostatic cancer, at least 2 months after the end of their radiation therapy. Participants will receive weekly treatments for 6 weeks.

The aims of the study are as follows:

Aim 1: To conduct a feasibility study to determine whether a 6-week SMT intervention can decrease CRF among prostate cancer survivors who have received radiation therapy and have CRF.

Aim 2: To determine whether the hypothesized decrease in CRF is due to SMT modulating the immune system of subjects with CRF. The researchers hypothesize that SMT will decrease plasma concentrations of IL-6 (a pro-inflammatory cytokine) more than LT and that the decrease in plasma IL-6 will mediate the decrease in fatigue as assessed with the MFI.

Aim 3: To determine whether SMT improves self-reported quality of life, depression, and anxiety more than LT, as assessed (respectively) by the Quality of Life, Enjoyment, and Satisfaction Questionnaire - short form (Q-LES-Q), the Quick Inventory of Depressive Symptoms - Self-Report (QIDS-SR), and the Generalized Anxiety Disorder 7-item (GAD-7) scale.

Aim 4: To evaluate the peripheral physiological changes associated with treatment of CRF. The researchers predict that treatment with SMT will cause a progressive increase in wearable measures of activity and step count, improved sleep quality (duration and latency), and decrease in pulse over 6 weeks when compared to baseline measures.

Aim 5: To determine if valid and useful tests of SMT effectiveness for treating CRF can be obtained through daily self-report ratings of fatigue and continuous monitoring of physiological signs. The researchers predict that SMT will cause a significant decrease in daily self-ratings of fatigue and mood when compared to baseline ratings and that the decreases in daily self-ratings of fatigue and mood observed with SMT will correlate with changes in Q-LES-Q, QIDS-SR, GAD-7 scores obtained at in-person visits as well as physiological signs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of prostate cancer
* At least 2 months after the end of radiation therapy
* Brief Fatigue Inventory (BFI) score of >25
* Satisfactory results of screening safety labs, serum testosterone test and drug test
* Ability to understand study procedures and to comply with them for the entire length of the study

Exclusion Criteria:

* Inability to lay supine for one hour at a time, given the nature of the massage intervention
* Actively suicidal or homicidal
* Medical conditions felt to be clinically contributing to fatigue based on the investigator's history, physical examination, and assessment: anemia (hemoglobin less than 10 g/dl), hypothyroidism (thyroid stimulating hormone greater than 4.6 microUnits per milliliter (mcU/mL)), uncontrolled pain, or medical problems associated with fatigue, including: chronic obstructive pulmonary disease, congestive heart failure, renal disease, hepatic dysfunction, autoimmune disease, neurological disorders such as multiple sclerosis or Parkinson's disease, and poorly controlled sleep apnea
* Medications felt to be clinically contributing to fatigue based on the investigator's history, physical examination, and assessment. Those may include: antidepressants, chronic use of long-acting anxiolytics or neuroleptics
* Treatment with high dose systemic corticosteroids or continuous use of other immunosuppressants within the past 30 days
* Unable to comply with the protocol for any reason
* Use of non-steroidal anti-inflammatory drugs; aspirin use is allowed but must be tracked
* Illicit drug use
* Shift work
* Currently dieting
* Excessive, regular use of alcohol (more than two 5 ounce glasses of wine or equivalents/day) or a history of binge drinking (more than 7 drinks/24 hour period) within the last 6 months
* Have used massage as a therapeutic modality (medical or psychological) at any point for the treatment of medical conditions
* Have massages on a regular basis, defined as receiving 4 or more massages per year for the last 5 years
* Currently employing any other complementary and alternative medicine (CAM) manual therapy and/or holistic therapies to treat a perceived health problem
* Unable to read and understand the informed consent document because of language difficulties
* Inability or unwillingness to give written informed consent

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Multidimensional Fatigue Inventory (MFI) score | Baseline, Week 6
  Multidimensional Fatigue Inventory (MFI) is a brief (20-item) self-report instrument that assesses 5 dimensions (subscales) of fatigue, including general fatigue, physical fatigue, mental fatigue, reduced activity, and reduced motivation. Respondents indicate their level of agreement with fatigue related statements on a 5 point scale ranging from "Yes, that is true" = 1 to "No that is not true" = 5. Possible scores for each subscale range from 4 (no fatigue) to 20 (maximum fatigue). The primary outcome measure for this study will be the total of four MFI subscales (general fatigue, physical fatigue, reduced activity, and reduced motivation).

SECONDARY OUTCOMES:
Change in Patient-Reported Outcome Measurement System (PROMIS) Fatigue Scale score | Baseline, Week 6
  The PROMIS Fatigue Scale is an 7-item self-report scale. Respondents indicate how tired they feel by answering fatigue related questions (such as "How often did you feel tired?") on a scale of 1 (never) to 5 (always). The summary score ranges from 7 to 35 with higher values equating to increased levels of fatigue.
Change in plasma IL-6 | Baseline, Week 6
  To examine the effects of SMT on the pro-inflammatory cytokine IL-6, blood will be drawn at each study visit and the plasma levels of IL-6 will be compared between prior to treatment and at treatment completion.
Change in Quality of Life, Enjoyment, and Satisfaction Questionnaire - short form (Q-LES-Q) score | Baseline, Week 6
  The Q-LES-Q short form is a 16-item, patient-administered instrument, which asks participants to rate their satisfaction with 13 specific areas of life, specifically, overall sense of well-being, medication, and overall life satisfaction and contentment during the past week. Responses are given on a 5-point scale where 1 = very poor and 5 = very good. Items 1-14 are added in order to obtain a summary score while the last two items are stand alone questions. Total scores range from 14 to 70 and higher scores indicate greater satisfaction with life.
Change in Quick Inventory of Depressive Symptomatology - Self-Report (QIDS-SR) score | Baseline, Week 6
  The QIDS-SR is a 16-item questionnaire covering nine diagnostic symptom domains that characterize a major depressive episode (sleep disturbance, sad mood, changes in appetite/weight, concentration, self-criticism, suicidal ideation, interest, energy/fatigue, and psychomotor agitation/retardation). The total score can range from 0 -27. A score of 1-5 equate to no depression while a score of 21-27 indicates very severe depression.
Change in Generalized Anxiety Disorder 7-item (GAD-7) Scale score | Baseline, Week 6
  The GAD-7 is a 7-item, well-validated patient self-report scale of anxiety. Participants respond to statements to indicate how often they have been bothered by specified symptoms of anxiety (such as "feeling nervous, anxious, or on edge). Response choices include 0 = not at all sure, 1 = several days, 2 = over half the days, and 3 = nearly every day. Total scores range from 0 to 21 with higher scores indicating increased anxiety.
Change in circadian variation of activity | Baseline, Week 6
  Activity level will be assessed by examining circadian variation (daily biologic cycles) of activity. Daily activity of each participant will be measured with a multisensor wristband device (Jawbone UP3). The device will collect data on activity levels and sleep metrics as participants wear the device throughout the study.
Change in step count | Baseline, Week 6
  The number of steps the participant takes each day will be measured with a multisensor wristband device (Jawbone UP3). The device will collect data on activity levels and sleep metrics as participants wear the device throughout the study.
Change in sleep duration | Baseline, Week 6
  The number of hours the participant sleeps each night will be measured with a multisensor wristband device (Jawbone UP3). The device will collect data on activity levels and sleep metrics as participants wear the device throughout the study.
Change in sleep latency | Baseline, Week 6
  The amount of time it takes for the participant to fall asleep will be measured with a multisensor wristband device (Jawbone UP3). The device will collect data on activity levels and sleep metrics as participants wear the device throughout the study.
Change in Automated Monitoring of Symptom Severity (AMoSS) survey score | Baseline, Week 6
  AMoSS is a smartphone app designed for longitudinal evaluation of mood states and sociability. Using this type of technology may help to better understand the day-to-day impact of SMT on the lives of cancer survivors with CRF, by means of a short pop-up survey that assesses sadness, anxiety, fatigue, irritability, and energy. Mood/fatigue will be assessed daily with reminders provided by the app via an alert.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rapaport, MD, Principal Investigator — Emory University
Locations (1):
- Executive Park 12, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided